CLINICAL TRIAL: NCT04219280
Title: Evaluating Assessment and Medication Treatment of ADHD in Children with Down Syndrome
Brief Title: Evaluating Treatment of ADHD in Children with Down Syndrome
Acronym: TEAM-DS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of California, Davis (Other); University of Pittsburgh Medical Center (Other); Boston Children's Hospital, Boston, MA, USA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-1016
Record Dates: First submitted 2019-12-31; First posted 2020-01-07 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Down Syndrome; ADHD
MeSH Terms: conditions — Down Syndrome; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Phase 1 is a Sequential model, Phase 2-3 is a Crossover model, Phase 4 is a Single-Group model.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quillivant XR (Active Comparator): Once-daily, long-lasting MPH solution with the following dosing schedules: 7.5mg/15mg/22.5mg/30mg for children 20-25kg 10mg/20mg/30mg/40mg for children 26-30kg 10mg/22mg/34mg/46mg for children > 30 mg
  Interventions: Drug: Quillivant XR
- Placebo (Placebo Comparator): Liquid-based suspension to match the color and banana-flavor of Quillivant XR.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quillivant XR — Long-lasting liquid solution of Quillivant XR.
  Arms: Quillivant XR
Drug: Placebo — Liquid solution to mimic the color and taste of Quillivant XR.
  Arms: Placebo

SUMMARY:
Children with Down syndrome (DS) have a 3-5 time greater prevalence of Attention Deficit Hyperactivity Disorder (ADHD) than typically developing (TD) children. Despite this higher risk of ADHD, rates of stimulant medication treatment are disproportionately low in children with DS+ADHD, even though stimulants are the most efficacious ADHD treatment and are recommended by consensus guidelines for use in children with intellectual disability and ADHD.

The investigators propose the first randomized clinical trial (RCT) of stimulant medication in children with DS+ADHD. This RCT may provide evidence regarding the short- and long-term safety and efficacy of stimulant use in children with DS+ADHD, both with and without CHD. All children enrolled in the study will complete a comprehensive assessment battery evaluating ADHD diagnostic criteria, as well as behavioral, cognitive, academic, and functional impairments.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a clinical trial of stimulant medication treatment (i.e., methylphenidate (MPH)) in children with DS+ADHD to determine methylphenidate's efficacy in remediating behavioral, cognitive, and functional impairments in children with DS+ADHD and to assess the short- and long-term safety of stimulant treatment in children with DS+ADHD with a specific focus on cardiac safety. It has the potential to significantly improve the outcomes of approximately 45,000 children with DS+ADHD nationwide.

To achieve this, 100 children with DS+ADHD, between the ages of 6.00-17.99 years, will be invited to participate in a clinical trial across four sites. Following pre-screening to determine study eligibility, children with DS+ADHD will be assessed at 13 different times points. The first pre-medication visit will include baseline intelligence, diagnostic, behavioral, cognitive, health, and functioning assessments. The second through sixth visits will begin Phase 1 of the clinical trial, and during this time, participants will begin the lowest dose of MPH and titrate incrementally upward per pediatric guidelines based on the participant's weight. Bieekly diagnostic and health assessments will be conducted to monitor the safety and efficacy of MPH during this phase. Further, this biweekly monitoring will ultimately guide the selection of the participant's optimal dose. At the seventh visit, participants will enter Phase 2 of the clinical trial where they will be randomized to receive an optimal dose of MPH (as determined by the assessments conducted throughout the titration phase) or the placebo. This visit will involve a repeat of most of the baseline measures. The eighth visit will initiate Phase 3 of the clinical trial in which participants will crossover to the study intervention not previously assigned during Phase 2. For example, a participant who was assigned his or her optimal dose during Phase 2 will receive the placebo during Phase 3, and vice versa. Further, this visit will involve a repeat of the assessments conducted during Phase 2 which allows each participants to serve as his or her own control, contributing data both while on an optimal dose of MPH and while on the placebo.

Prior to commencing Phase 4, MPH non-responders or placebo responders will be removed from the study and referred for non-study (clinical) treatment. Participants for whom MPH is judged to be effective and tolerable based on clinician ratings and parent/teacher reports will be invited to undergo an open label trial with their optimal MPH dose for a four-month maintenance period. During this phase, participants will undergo monthly diagnostic and health assessments to monitor the safety and efficacy of his or her optimal dose of MPH. The final visit (week 30) will include diagnostic, behavioral, cognitive, functioning, and health assessments to evaluate change across time.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, between the ages of 6.00-17.99 years at the time of consent.
* Able to take oral (liquid) medication.
* English is primary language.
* Meets criteria for ADHD (hyperactivity, inattention, or combined) on the KSADS
* Meets criteria for ADHD (hyperactivity, inattention, or combined) on the Vanderbilt (historically or currently, as indicated by a teacher/professional)

Exclusion Criteria:

* Current use of ADHD stimulant or non-stimulant medication and unwilling to discontinue for >/= 3 days prior to starting the study.
* Children with psychoses or bipolar disorder based on diagnostic interview with the parent.
* Organic Brain Injury: Children must not have a history of head trauma with loss of consciousness, epilepsy, or any other organic disorder that could possibly affect brain function.
* Specific heart conditions including the following:

  1. QTc on baseline ECG>470ms or QTC > 500 in patients with repaired CHD, as determined by ECG
  2. Brugada pattern, as determined by ECG
  3. Baseline heart rate or systolic blood pressure > 2 SD above mean for age as determined by medical examination.
  4. 2nd or 3rd degree AV block, as determined by ECG
  5. History of aborted sudden cardiac death or unexplained syncope as determined by medical history
  6. History of a single ventricle as determined by medical history
  7. Valvular regurgitation or stenosis > mild, as determined by ECHO
  8. Moderate or greater ventricular dysfunction, as determined by ECHO
  9. Pulmonary hypertension, defined as right ventricular pressure >33% systemic pressure or septal position consistent with >mild right ventricular hypertension, as determined by ECHO
  10. Use of a pacemaker as determined by medical history
  11. Wolff Parkinson White/pre-ventricular excitation, as determined by ECG
  12. Atrial, junctional, or ventricular tachyarrhythmia, as determined by ECG
  13. Frequent premature ventricular contractions (PVCs) or premature atrial contractions (PACs), as determined by ECG
  14. Abnormal T waves with inversion in V5 and/or V6, bizarre T wave morphology, notched biphasic T waves, or ST segment depression suggesting ischemia or inflammation, as determined by ECG
  15. Moderate or larger atrial septal defect, as determined by ECHO
  16. Ventricular septal defect > small by ECHO
  17. Valvar stenosis > mild by ECHO
  18. Aortic root dilation > 2SD above mean by ECHO.
* If participants meet any of the following heart conditions, they must be evaluated for the study by a cardiologist before beginning:

  1. Right ventricular enlargement/right axis deviation, as determined by ECG
  2. Intraventricular conduction delay >120ms in child >12 years old or >100ms in child <8 years old, as determined by ECG
  3. Right or left bundle branch block, as determined by ECG
* Treatment with a monoamine oxidase inhibitor (MAOI) or use of an MAOI within 14 days.
* Active titration of non-ADHD, non-MAO psychotropic medication. Stable use of non-ADHD, non-MAO psychotropic medication, defined by no dose changes for >/= 4 weeks before starting the study medication trial, will be allowed.
* Known hypersensitivity or allergic reactions to methylphenidate or product components such as banana (due to bananas serving as flavoring in the formulation of the project's study interventions - Quillivant XR and the placebo).
* Severe Obstructive Sleep Apnea (OSA) as rated by McGill index of 4
* Pregnancy. (Since there is limited information regarding the safety of Quillivant XR during pregnancy, a pregnancy test will be conducted at the medical screen for female participants who have commenced the menstrual cycle. If pregnancy is indicated, the participant will be excluded from the study as a precautionary measure).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean magnitude of change in ADHD Symptoms as measured by parent and teacher report on the Vanderbilt ADHD Parent and Teacher Rating Scales, compared to placebo, during the optimal MPH dosage period. [ Time Frame: Phase 2, Phase 3 ] | Baseline, Weeks 2-14, Weeks 18, 22, 26, and 30
  A 49-item parent-report measure used to assess parent and teacher perceptions of youth's school and social functioning. The first 47 items assess symptoms of inattention, hyperactivity, combined inattention and hyperactivity, oppositional-defiant disorder, conduct disorder, and anxiety/depression. These items are scored on a 0-3 scale (0 = Never; 1 = Occasionally; 2 = Often; 3 = Very Often). The next two items measure impairment in performance and are scored on a 1-5 scale (1 = Above Average; 3 = Average; 5 = Problematic). For both sub-scales, lower scores mean better outcomes. Data will be entered into SPSS and used as a diagnostic outcome measure.
Mean magnitude of change in Emotion Regulation as measured by parent and teacher report on the BRIEF2, compared to placebo, during the optimal MPH dosage period. [ Time Frame: Phase 2, Phase 3 ] | Baseline, Week 12, Week 14, and Week 30
  A 63-item parent and teacher rating scale used to assess everyday skills measuring executive functioning, including inhibition, shifting attention, emotional control, initiating tasks, problem solving, working memory, and monitoring activities. All 63-items are scored on a 3-item scale (N = never, S = Sometimes, O = Often). Scoring is performed through a software which generates T-scores for 13 sub-scales, with borderline and clinical ranges identified. Lower scores on this measure indicate better outcomes. Data will be entered into SPSS and used as a behavioral outcome measure.

SECONDARY OUTCOMES:
Mean magnitude change in Externalizing Behaviors as measured by parent and teacher report on the Achenbach Child Behavior Checklist (CBCL/TRF), compared to placebo, during the optimal MPH dosage period. [ Time Frame: Phase 2, Phase 3 ] | Baseline, Week 12, Week 14, and Week 30
  A 113-item rating scale used to obtain parent and teacher ratings of problem behaviors, in addition to descriptions of a child's strengths and challenges. All items are scored on a 0-2 scale (0 = Not True; 1 = Somewhat True or Sometimes True; 2 = Very True or Often True). T-scores for 8 sub-scales with borderline and clinical ranges are generated and identified through a scoring software, and lower scores on this measure indicate better outcomes. Data will be entered into SPSS and used as a behavioral outcome measure.
Mean magnitude of change in Behavior Regulation as measured by parent and teacher report on the BRIEF2, compared to placebo, during the optimal MPH dosage period. [ Time Frame: Phase 2, Phase 3 ] | Baseline, Week 12, Week 14, and Week 30
  A 63-item parent and teacher rating scale used to assess everyday skills measuring executive functioning, including inhibition, shifting attention, emotional control, initiating tasks, problem solving, working memory, and monitoring activities. All 63-items are scored on a 3-item scale (N = never, S = Sometimes, O = Often). Scoring is performed through a software which generates T-scores for 13 sub-scales, with borderline and clinical ranges identified. Lower scores on this measure indicate better outcomes. Data will be entered into SPSS and used as a behavioral outcome measure.
Frequency of clinically significant physician-collected cardiac occurrences on MPH - clinically significant change from baseline in ECG findings during the during the MPH titration trial [Phase 1] and the optimal MPH dosage maintenance period [Phase 4]. | Baseline, Week 8, Week 10, Week 22, and Week 30
  An ECG will be acquired at standard amplitude and speed (10mm/mV and 25mm/sec), and an electrophysiologist will inspect the recorded ECG for satisfactory quality and findings. The electrodes and lead wires will be applied to the extremities and chest with proper lead placement.The ECG readings will be used to assess the cardiovascular safety of stimulant medication treatment among the participants. Data will be reviewed by a cardiologist, and entered into SPSS to serve as a safety outcome measure.
Frequency of clinically significant cardiac occurrences on MPH- clinically significant changes for Heart Rate (HR) during the MPH titration trial [Phase 1] and the MPH dosage maintenance period [Phase 4]. | Baseline, Weeks 2-14, Weeks 18, 22, 26, and 30
  HR will be assessed and collected by trained study staff and clinically significant changes will be tracked and assessed based on the participant's age.
Frequency of clinically significant cardiac occurrences on MPH- clinically significant changes for Blood Pressure (BP) during the MPH titration trial [Phase 1] and the MPH dosage maintenance period [Phase 4]. | Baseline, Weeks 2-14, Weeks 18, 22, 26, and 30
  BP measurement will be acquired by trained study staff or medical staff and clinically significant changes will be tracked and assessed based on the participant's age and height.
Mean magnitude of change in Heart Rate (HR) compared to participants' pre-trial baseline, on maximum dosage of MPH received during the MPH titration trial [Phase 1] and during the optimal MPH dosage maintenance period [Phase 4]. | Baseline, Weeks 2-14, Weeks 18, 22, 26, and 30
  HR will be acquired at each visit and compared to baseline measurements based on participant's age.
Mean magnitude of change in Systolic Blood Pressure (SBP) compared to participants' pre-trial baseline, on maximum dosage of MPH received during the MPH titration trial [Phase 1] and during the optimal MPH dosage maintenance period [Phase 4]. | Baseline, Weeks 2-14, Weeks 18, 22, 26, and 30
  SBP will be acquired at each visit and compared to baseline measurements based on participant's age and height.
Mean magnitude of change in Diastolic Blood Pressure (DBP) compared to participants' pre-trial baseline, on maximum dosage of MPH received during the MPH titration trial [Phase 1] and during the optimal MPH dosage maintenance period [Phase 4]. | Baseline, Weeks 2-14, Weeks 18, 22, 26, and 30
  DBP will be acquired at each visit and compared to baseline measurement based on participant's age and height.
Frequency of parent-rated MPH side effects | Baseline, Weeks 2-14, Weeks 18, 22, 26, and 30
  A 19-item parent rating scale used to assess known side effects will be administered at each visit using a 4-item scale (0-None, 1-Mild, 2-Moderate, 3-Severe). A medical interview will be conducted to discuss side effects outside of the scope of this measurement and any unexpected or unrelated side effects or adverse events,

CONTACTS AND LOCATIONS:
Overall Officials: Anna Esbensen, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Tanya Froehlich, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Kathleen Angkustsiri, MD, Principal Investigator — University of California Davis MIND Institute; Benjamin Handen, MD, Principal Investigator — University of Pittsburgh Medical Center; Sabrina Sargado, MD, Principal Investigator — Boston Children's Hospital
Locations (4):
- United States (4):
  - University of California Davis MIND Institute, Sacramento, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The research team will enter information in the clinical trial record at least once per year, and will enter the results of the primary outcomes within one year of the completion of the trial.
  The dataset generated and shared will include de-identified demographic information, parent- and teacher-rating scales, side effects and vital signs, cardiac monitoring, and blinded clinical global impressions. The dataset will include all composite variables and scores, with no identifying information included. The data and associated documentation will be made available to users only under a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Due to the nature of data collection in a blinded randomized clinical trial, data will be made available upon completion of sampling and primary analyses. Data will also be archived in accordance with the scientific journals in which reports from the project are published.
  Prior to publication, findings from the project will be shared broadly at conferences attended by professionals doing intervention work with the children with intellectual and developmental disabilities, and at scientific meetings attended by researchers focused on intellectual and developmental disabilities.
Access Criteria: Data will be shared at the completion of the project according to any and all NIH guidelines. Furthermore, data may be shared with colleagues at other sites in the future, but only under conditions specified by the IRBs at the participating universities and research sites, and in a manner consistent with written informed consent provided by the participants.